CLINICAL TRIAL: NCT06143891
Title: A Randomized, Double-blind, Multicenter, Phase 3 Study to Evaluate Efficacy and Safety of Belumosudil in Combination With Corticosteroids Versus Placebo in Combination With Corticosteroids in Participants at Least 12 Years of Age With Newly Diagnosed Chronic Graft Versus Host Disease (cGVHD)
Brief Title: A Study to Test an Oral Medicine, Belumosudil, in Combination With Corticosteroids in Participants at Least 12 Years of Age With Newly Diagnosed Chronic Graft Versus Host Disease.
Acronym: ROCKnrol-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17757; 2023-505394-32 (Registry Identifier: CTIS); U1111-1280-4918 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil; KD025; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belumosudil (Experimental): Participants will receive belumosudil 200 mg tablets per os(PO) once daily (QD) per 28-day cycles starting on Day 1 until discontinuation criteria are met or until end of study
  Note: 200mg two times a day (BID) is used in some cases, when the subject is taking a proton pump inhibitor or a strong CYP3A4 inducer)
  Interventions: Drug: Belumosudil; Drug: Prednisone; Drug: Prednisolone
- Placebo (Placebo Comparator): Participants will receive matching placebo tablets PO QD per 28-day cycles starting on Day 1 until discontinuation criteria are met or until end of study
  Interventions: Drug: Placebo; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form:Tablet-Route of administration:oral
  Other Names: SAR445761/ KD025; REZUROCK
  Arms: Belumosudil
Drug: Placebo — Pharmaceutical form:Table-Route of administration:oral
  Arms: Placebo
Drug: Prednisone — Pharmaceutical form:Tablet-Route of administration:oral
Drug: Prednisolone — Pharmaceutical form:Tablet-Route of administration:oral

SUMMARY:
This is a parallel, Phase 3, two-arm study for the treatment of newly diagnosed moderate or severe chronic GVHD.

The study duration for a participant includes up to 4 weeks for screening; a treatment period until clinically meaningful cGVHD progression (defined as progression requiring addition of new systemic treatment for cGVHD), relapse/recurrence of the underlying disease, participant starts new systemic treatment for cGVHD or experiences an unacceptable toxicity, at the request of the participants or the investigators, or until the end of study is reached, whichever comes first; at least 30 days follow-up of adverse events (AEs) after the last dose until resolution or stabilization, if applicable; and long-term follow-up until death or study close-out, whichever comes first.

DETAILED DESCRIPTION:
Up to 2.5 years

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 12 years of age inclusive, at the time of signing the informed consent
* Participants who have undergone allogenic HCT with newly diagnosed moderate to severe cGVHD according to NIH consensus diagnosis and staging criteria (2014)
* Participants who require systemic treatment with corticosteroids for cGVHD
* Participants who have not received any prior systemic treatment for cGVHD (including ECP)
* If participants are receiving other immunosuppressive agents for the prophylaxis or treatment of acute GVHD, the dose should be under the threshold pre-defined in protocol
* For adult participants, the body weight should be ≥40 kg. For adolescent participants, the body weight should be ≥30 kg
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Participants or their legally authorized representative must be capable of giving signed informed consent

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical conditions

* Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of progressive or relapsed underlying disease after the most recent allogeneic HCT
* Post-transplant lymphoproliferative disease within 4 weeks prior to randomization
* Female participants who are pregnant or breastfeeding
* Unable to tolerate a prednisone equivalent dose of corticosteroids ≥ 1 mg/kg/day Prior/concomitant therapy
* Participant has had previous exposure to belumosudil.
* Received any previous systemic treatment for cGVHD with the following exception: Corticosteroids for cGVHD received within 7 days prior to the planned administration of IMP only if in the interest of participant.

Prior/concurrent clinical study experience

* Received any investigational agents, or any investigational device or procedure, or prohibited therapy for this study within 28 days or 5 elimination half-lives prior to randomization, whichever is longer Diagnostic assessments
* Karnofsky (if aged ≥16 years)/Lansky (if aged <16 years) Performance Score of < 60
* Platelets <25 x 109/L. Platelet transfusion is not allowed within 3 days before the screening hematological test
* Absolute neutrophil count (ANC) <0.5 x 109/L. The use of granulocyte-colony stimulating factor (G-CSF) is not allowed to reach this level during screening
* Estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73 m2 using the MDRD-4 variable formula (if aged ≥18 years) or using the Bedside Schwartz formula (if aged <18 years)
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3 x ULN without liver cGVHD or>5 × ULN with liver) cGVHD
* Total bilirubin >1.5 × (ULN) (>3 × ULN if Gilbert syndrome)
* Participant has forced expiratory volume in 1 second (FEV1) of predicted ≤39% or has lung score of 3 according to NIH consensus diagnostic and staging criteria (2014)
* History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study (such as malabsorption syndromes, poorly controlled psychiatric disease or coronary artery disease)
* Known history of human immunodeficiency virus (HIV)
* Active viral disease including hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Active uncontrolled cytomegalovirus (CMV) and Epstein-Barr virus (EBV) infection. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of infection worsening are present according to Investigator's judgement
* Diagnosed or treated for another malignancy other than the underlying disease allogeneic HCT was indicated for, within 3 years prior to randomization with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in-situ malignancy, or low risk prostate cancer after curative therapy
* Unable to swallow tablets
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures
* Any active, uncontrolled infections assessed to be clinically significant by the Investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2028-09-29 (Estimated); Study Completion 2028-09-29 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | Until the end of the study (up to 2.5 years since first patient in).
  From the date of randomization to the date of any predefined event, whichever occurs first

SECONDARY OUTCOMES:
Modified Lee Symptom Scale (mLSS) | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants who achieve a clinically relevant reduction in mLSS of at least 6 points from baseline (Only in participants at least 18 years of age)
Durable overall response rate | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants who achieve an overall response (PR or CR) as per 2014 NIH consensus response criteria by 48 weeks and maintained the response for a duration of at least 6 months
Rate of corticosteroid withdrawal | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants who successfully discontinue all systemic corticosteroids for cGVHD for at least 30 days before the occurrence of cGVHD progression, or start of a new systemic treatment for cGVHD, relapse or recurrence of the underlying disease, or unacceptable toxicity
Overall response rate (ORR) | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants who achieve an overall response (CR or PR) as per 2014 NIH consensus response criteria at any time before the start of new systemic treatment for cGVHD
ORR by 24 weeks | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants who achieve an overall response (CR or PR) as per 2014 NIH consensus response criteria by 24 weeks (Cycle 7 Day 1) before the start of new systemic treatment for cGVHD
Duration of response (DOR) | Until the end of the study (up to 2.5 years since first patient in).
  Time from the date of the first response to the date of cGVHD progression, start of new systemic treatment for cGVHD, or death, whichever occurs first. DOR is determined only for participants who achieved overall response (PR or CR) as per 2014 NIH consensus response criteria
Dose reduction in corticosteroid | Until the end of the study (up to 2.5 years since first patient in).
  Proportion of participants with a reduction in daily corticosteroid dose
Failure Free Survival (FFS) | Until the end of the study (up to 2.5 years since first patient in).
  Failure Free Survival (FFS) is defined as the time from the date of randomization to the date of start of a new systemic treatment for cGVHD, relapse or recurrence of the underlying disease, or death, whichever occurs first.
Change in patient reported outcome (PRO) | Until the end of the study (up to 2.5 years since first patient in).
  Change from baseline in Patient-Reported Outcomes Measurement Information System Global Health (PROMIS-GH) (Only in participants at least 18 years of age) and the European Quality of Life Group Questionnaire with 5 Dimensions and 5 Levels (EQ5D5L)
Number of participants with treatment-emergent adverse events [TEAEs], serious TEAEs, and adverse events of special interest (AESIs) | Until the end of the study (up to 2.5 years since first patient in).
Overall survival | Until the end of the study (up to 2.5 years since first patient in).
  The time from the date of randomization to the date of death due to any cause
Time to response (TTR) | Until the end of study (up to 2.5 years since first patient in)
  Time to Response is defined as the time from randomization to the date the patient has first response (CR or PR).
Response by organ | Until the end of study (up to 2.5 years since first patient in)
  Proportion of participants who achieve CR or PR as per NIH consensus response criteria (2014) at any time point in each involved organ and before the start of a new systemic therapy for cGVHD.

CONTACTS AND LOCATIONS:
Locations (151):
- United States (24):
  - University of Arkansas for Medical Sciences-Site Number : 8400019, Little Rock, Arkansas
  - City of Hope National Medical Center- Site Number : 8400001, Duarte, California
  - University of California San Francisco - Parnassus Heights- Site Number : 8400035, San Francisco, California
  - AdventHealth Orlando- Site Number : 8400023, Orlando, Florida
  - The Hope Clinic of Emory University- Site Number : 8400020, Decatur, Georgia
  - Northwestern University- Site Number : 8400017, Chicago, Illinois
  - Indiana University Health University Hospital- Site Number : 8400006, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center- Site Number : 8400024, Lexington, Kentucky
  - Johns Hopkins Hospital- Site Number : 8400033, Baltimore, Maryland
  - Dana Farber Cancer Institute Site Number : 8400005, Boston, Massachusetts
  - Karmanos Cancer Institute - Detroit- Site Number : 8400013, Detroit, Michigan
  - UNC Children's Hospital- Site Number : 8400025, Chapel Hill, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center - Winston-Salem - Medical Center Boulevard- Site Number : 8400007, Winston-Salem, North Carolina
  - Oncology Hematology Care - Kenwood- Site Number : 8400030, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center (OSUCCC) - The James Cancer Hospital and Solove Research Institute- Site Number : 8400026, Columbus, Ohio
  - Oregon Health and Science University- Site Number : 8400027, Portland, Oregon
  - UPMC Hillman Cancer Center- Site Number : 8400008, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute Site Number : 8400003, Nashville, Tennessee
  - St. David's South Austin Medical Center- Site Number : 8400002, Austin, Texas
  - Texas Oncology - Dallas - Worth Street- Site Number : 8400010, Dallas, Texas
  - Texas Transplant Institute - Methodist Hospital- Site Number : 8400037, San Antonio, Texas
  - University of Virginia Comprehensive Cancer Center-Site Number : 8400031, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center- Site Number : 8400004, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center-Site Number : 8400029, Madison, Wisconsin
- Argentina (6):
  - Investigational Site Number : 0320006, Pilar, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Córdoba
- Australia (4):
  - Investigational Site Number : 0360005, Westmead, New South Wales
  - Investigational Site Number : 0360003, Brisbane, Queensland
  - Investigational Site Number : 0360001, Melbourne, Victoria
  - Investigational Site Number : 0360004, Murdoch, Western Australia
- Austria (3):
  - Investigational Site Number : 0400003, Graz
  - Investigational Site Number : 0400001, Linz
  - Investigational Site Number : 0400004, Vienna
- Belgium (6):
  - Cliniques Universitaires St. Luc-Investigational Site Number : 0560005, Woluwe, Brussels Capital
  - UZ Leuven-Investigational Site Number : 0560001, Leuven, Vlaams-Brabant
  - Investigational Site Number : 0560006, Bruges
  - UZ Gent-Investigational Site Number : 0560003, Ghent
  - CHU de Liège-Investigational Site Number : 0560004, Liège
  - AZ Delta-Investigational Site Number : 0560002, Roeselare
- Brazil (5):
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760008, Curitiba, Paraná
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto- Site Number : 0760006, São José do Rio Preto, São Paulo
  - INCA - Hospital do Câncer - Rio de Janeiro - Praça Da Cruz Vermelha- Site Number : 0760007, Rio de Janeiro
  - Hospital das Clinicas FMUSP- Site Number : 0760004, São Paulo
  - Hospital Israelita Albert Einstein- Site Number : 0760003, São Paulo
- Canada (6):
  - Investigational Site Number : 1240007, Calgary, Alberta
  - Investigational Site Number : 1240005, Toronto, Ontario
  - Hôpital Maisonneuve Rosemont-Investigational Site Number : 1240001, Montreal, Quebec
  - CHU Sainte-Justine-Site Number : 1240003, Montreal, Quebec
  - Investigational Site Number : 1240002, Montreal, Quebec
  - Investigational Site Number : 1240008, Saskatoon, Saskatchewan
- China (16):
  - Investigational Site Number : 1560019, Beijing
  - Investigational Site Number : 1560012, Changchun
  - Investigational Site Number : 1560010, Changsha
  - Investigational Site Number : 1560011, Fuzhou
  - Investigational Site Number : 1560005, Guangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560014, Hefei
  - Investigational Site Number : 1560008, Jinan
  - Investigational Site Number : 1560007, Jinan
  - Investigational Site Number : 1560001, Suzhou
  - Investigational Site Number : 1560006, Suzhou
  - Investigational Site Number : 1560003, Tianjin
  - Investigational Site Number : 1560004, Tianjin
  - Investigational Site Number : 1560013, Wuhan
  - Investigational Site Number : 1560015, Wuhan
  - Investigational Site Number : 1560009, Zhengzhou
- Czechia (4):
  - Interni hematologicka a onkologicka klinika Fakultni nemocnice Brno-Site Number : 2030003, Brno
  - IV. Interni hematologicka klinika, Fakultni nemocnice Hradec Kralove-Site Number : 2030002, Hradec Králové
  - Klinika hematoonkologie, Fakultni nemocnice Ostrava-Site Number : 2030001, Ostrava
  - Ustav hematologie a krevni transfuze-Site Number : 2030004, Prague
- Denmark (3):
  - Rigshospitalet Copenhagen University Hospital-Investigational Site Number : 2080002, Copenhagen, Capital
  - Odense University Hospital-Investigational Site Number : 2080003, Odense, Funen
  - Department of hematology-Investigational Site Number : 2080001, Aarhus, Jutland
- France (8):
  - Institut Paoli Calmettes-Investigational Site Number : 2500004, Marseille
  - CHU Hotel Dieu-Investigational Site Number : 2500005, Nantes
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500001, Paris
  - CHU Bordeaux-Hôpital Haut-Lévêque-Investigational Site Number : 2500002, Pessac
  - Hôpital Lyon Sud-Investigational Site Number : 2500007, Pierre-Bénite
  - Hôpital Pontchaillou - CHU de Rennes-Investigational Site Number : 2500008, Rennes
  - Investigational Site Number : 2500006, Vandœuvre-lès-Nancy
- Germany (9):
  - Investigational Site Number : 2760007, Berlin
  - Investigational Site Number : 2760003, Cologne
  - Investigational Site Number : 2760001, Dresden
  - Investigational Site Number : 2760005, Freiburg im Breisgau
  - Investigational Site Number : 2760002, Hamburg
  - Investigational Site Number : 2760010, Kiel
  - Investigational Site Number : 2760009, Münster
  - Investigational Site Number : 2760006, Regensburg
  - Investigational Site Number : 2760008, Tübingen
- Greece (2):
  - Nosokomeio Paidon I Agia Sofia-Site Number : 3000002, Athens
  - General Hospital of Thessaloniki "George Papanikolaou"-Site Number : 3000001, Thessaloniki
- Investigational Site Number : 3440001, Pok Fu Lam, Hong Kong
- Israel (6):
  - Investigational Site Number : 3760002, Haifa
  - Investigational Site Number : 3760005, Jerusalem
  - Investigational Site Number : 3760006, Petah Tikva
  - Investigational Site Number : 3760003, Ramat Gan
  - Investigational Site Number : 3760004, Ramat Gan
  - Investigational Site Number : 3760001, Tel Aviv
- Italy (12):
  - Investigational Site Number : 3800012, Torette, Ancona
  - Investigational Site Number : 3800005, Genoa, Genova
  - Investigational Site Number : 3800009, Milan, Milano
  - Investigational Site Number : 3800002, Rozzano, Milano
  - Investigational Site Number : 3800001, Rome, Roma
  - Investigational Site Number : 3800007, Turin, Torino
  - Investigational Site Number : 3800003, Bergamo
  - Investigational Site Number : 3800004, Bologna
  - Investigational Site Number : 3800011, Pavia
  - Investigational Site Number : 3800010, Perugia
  - Investigational Site Number : 3800006, Reggio Calabria
  - Investigational Site Number : 3800008, Udine
- Netherlands (4):
  - Amsterdam Universitair Medisch Centrum-Site Number : 5280005, Amsterdam
  - Investigational Site Number : 5280003, Groningen
  - Investigational Site Number : 5280002, Rotterdam
  - Investigational Site Number : 5280001, Utrecht
- Poland (2):
  - Investigational Site Number : 6160001, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160008, Szczecin
- Portugal (2):
  - Investigational Site Number : 6200003, Lisbon
  - Investigational Site Number : 6200002, Lisbon
- South Korea (4):
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
- Spain (10):
  - Investigational Site Number : 7240011, Santander, Cantabria
  - Investigational Site Number : 7240005, Barcelona, Catalunya [Cataluña]
  - ICO Institut Català d'Oncologia-Site Number : 7240006, Barcelona, Catalunya [Cataluña]
  - Investigational Site Number : 7240004, Madrid
  - Hospital Niño Jesús-Site Number : 7240002, Madrid
  - Hospital Regional Universitarioa de Malaga-Site Number : 7240003, Málaga
  - Hospital Universitario de Salamanca-Site Number : 7240007, Salamanca
  - Hospital Universitario Virgen del Rocío.-Site Number : 7240008, Seville
  - Investigational Site Number : 7240012, Valencia
  - Hospital Universitari i Politècnic La Fe-Site Number : 7240001, Valencia
- Sweden (3):
  - Investigational Site Number : 7520003, Gothenburg
  - Investigational Site Number : 7520001, Huddinge
  - Investigational Site Number : 7520002, Lund
- Turkey (Türkiye) (6):
  - Investigational Site Number : 7920006, Adana
  - Investigational Site Number : 7920002, Ankara
  - Investigational Site Number : 7920004, Ankara
  - Investigational Site Number : 7920001, Ankara
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920003, Izmir
- United Kingdom (5):
  - Investigational Site Number : 8260006, Cardiff, Cardiff [Caerdydd Gb-crd]
  - Investigational Site Number : 8260002, London, London, City of
  - Investigational Site Number : 8260003, Leeds
  - Investigational Site Number : 8260001, Manchester
  - Investigational Site Number : 8260004, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17757 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25529&tenant=MT_SNY_9011